CLINICAL TRIAL: NCT00299598
Title: phase2 Safety and Efficacy of Antibacterial Nano Particles Incorporated in Dental Composite.
Brief Title: Clinical Study of Antibacterial Nanoparticles Incorporated in Composite Restorations
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: 191060HMO-CTIL
Record Dates: First submitted 2006-03-05; First posted 2006-03-07 (Estimated); Last update posted 2010-01-06 (Estimated); Status verified 2009-10

CONDITIONS: Oral Health
Keywords: antibacterial; composite; polyethylenimine; nanoparticle

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

INTERVENTIONS:
Device: alkylated polyethylenimine nanoparticles antibacterial evaluation

SUMMARY:
Resin composites withholding antibacterial properties may be useful in preventing recurrent caries. Covalently attached antibacterial polymers are a possible solution.This in vivo study would evaluated the antibacterial effect of alkylated polyethylenimine nanoparticles incorporated into flowable and hybrid composite resin disks embedded in a palatal removable appliance.The disks would be in close contact with the palate in order to check for contact mucosities. disks on the side facing the Tongue would be evaluated for their antibacterial potency with confocal laser scanning microscopy.

DETAILED DESCRIPTION:
Composite resin materials are widely used in the dental clinic for replacement of hard tissues. Although the mechanical properties and wear resistance of these materials have been improved substantially, their antibacterial properties are still limited. These resin-based materials accumulate more dental plaque than other restorative materials both in vitro, and in vivo, which may result in secondary caries. A number of reports described experiments in which composite resins were impregnated with antibacterial agents such as antibiotics, silver ions, iodine and quaternary ammonium compounds, and gradually released them. However, release of antibacterial agents into the surrounding milieu at various releasing rates had several disadvantages: a decrease in the mechanical properties of the carrier material over time, short-term effectiveness, and possible toxicity if the release is not properly controlled. As compared with conventional antibacterial agents of low molecular weight, the advantage of polymeric antibacterial agents is that they are nonvolatile, chemically stable, can be chemically bound within the polymer carrier via active groups for improved integration in the composite, and are difficult to penetrate through the skin. It has been reported that polycations exhibit antibacterial properties, i.e. interact with and disrupt bacterial cell membranes. A number of polymers with antibacterial properties were developed for this purpose, including soluble and insoluble pyridinium-type polymers involved in surface coating. Several reports have described incorporation of a methacryloyloxydodecylpydidinium bromide (MDPB) monomer in composite resins that showed no release of the incorporated monomer but still exhibited antibacterial properties. The objective of this study is to evaluate clinically the safety and efficacy of alkylated polyethylenimine (PEI) nanoparticles in composite resin restorative materials . In an in vitro study, addition of a small percent (1% w/w) of nanoparticles did not affect significantly the flexural strength of the commercial materials. The mechanical properties of the new composites were close to those of the original composite, but exerted a strong antibacterial activity upon contact that lasted for at least six months.

methods:alkylated polyethylenimine (PEI) nanoparticles added (1% w/w)to hybrid composite resin disks embedded in a palatal removable appliance.The disks would be in close contact with the palate in order to check for contact mucosities. disks on the side facing the Tongue would be evaluated for their antibacterial potency with confocal laser scanning microscopy.

ELIGIBILITY:
Inclusion Criteria:healthy

* must be able to wear upper removable appliance

Exclusion Criteria:

* gag reflex
* infectious disease

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: personal of Hadassah MO
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2006-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ervin I Weiss, DMD, Study Chair — Hadassah Medical Organization; Avi Domb, Phd, Study Director — Hebrew University of Jerusalem; Michael M Perez Davidi, DMD, Principal Investigator — Hadssah Medical Orgenization; Nurit Beyth, DMD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Result] Matalon S, Slutzky H, Weiss EI. Surface antibacterial properties of packable resin composites: part I. Quintessence Int. 2004 Mar;35(3):189-93. PMID 15119676
- See also: Michael Perez Davidi — http://www.mypd.co.il